CLINICAL TRIAL: NCT05355337
Title: Adjunctive Treatment With Pramipexole for Anhedonic Depression Symptoms in Depression - PRIME-PRAXOL
Brief Title: Pramipexole for Anhedonic Depression
Acronym: PRIME-PRAXOL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-06876-01; 2022-001563-26 (EudraCT Number)
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Disorders Mood; Anhedonia; Depression
Keywords: Pramipexole
MeSH Terms: conditions — Mood Disorders; Anhedonia; Depression | interventions — Pramipexole

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled with two arms plus one arm of healthy controls with no intervention
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pramipexole (Active Comparator): Pramipexole prolonged-release tablet, 0.26 mg base to 3.15 mg base / day for 9 weeks (individually varying dose titrating during these weeks).
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Tablets in appearance identical to the active comparator tablets, but without the the active substance (pramipexole).
  Interventions: Drug: Placebo
- Healthy controls (No Intervention): 40 healthy controls who will carry out blood sampling, lumbar puncture and fMRI according to the same protocol as the depressed patients.

INTERVENTIONS:
Drug: Pramipexole — 9 weeks of treatment with Pramipexole
  Arms: Pramipexole
Drug: Placebo — 9 weeks of treatment with Placebo
  Arms: Placebo

SUMMARY:
The heterogeneity of depression suggests that several different neurocircuits and pathophysiological mechanisms are involved. Anhedonia - the inability to experience pleasure from, or the lack of motivation to carry out, usually enjoyable activities - is a promising endophenotype within the depression spectrum, with a distinct pathophysiology involving dopaminergic mesolimbic projections. Anhedonia is common in depression and associated with treatment resistance. Pramipexole, an agonist to the dopamine -receptor 3, is an established treatment of Parkinson's disease. Based on its mechanism of action, pramipexole might be efficacious in a subtype of depression characterized by anhedonia and lack of motivation - symptoms linked to dopaminergic hypofunction. This is supported by animal data, clinical experience, and recent pilot study data, but randomized controlled trials (RCTs) are lacking. In this double-blind placebo-controlled RCT the anti-anhedonic and antidepressant effects of add-on pramipexole will be tested, using an "enriched population study design" including only depressed patients with significant anhedonia. To better understand the neurobiology of anhedonia in depression and to identify treatment predictors, simultaneous assessments of anhedonia-related neurocircuitry using (f)MRI will be done, and anhedonia-related biomarkers in blood and cerebrospinal fluid analyzed. The aim of the study is to confirm the efficacy of pramipexole in this depression subtype, which would be an important step towards personalized medicine in psychiatry.

DETAILED DESCRIPTION:
This is a randomized, double-blind drug trial in which 80 patients are included and treated with adjuvant pramipexole or placebo for 9 weeks. The treatment trial will be supplemented by two sub-trials with fMRI examination and lumbar puncture in research subjects who wish to participate (not mandatory for participation in the main trial).

The aim of the project is to administer pramipexole as an adjuvant to ongoing antidepressant treatment of patients with affective disorders with a symptom profile characterized by anhedonia. This trial may fill an important knowledge gap through i) the inclusion of depressive patients with significant anhedonia symptoms regardless of baseline diagnosis, ii) the use anhedonia symptoms as the primary outcome measure, iii) the use higher doses of pramipexole compared to previous studies and iv) the use of fMRI and biomarkers to predict treatment response in the future. In order to achieve a higher dosage and sufficient treatment effect compared to previously, and avoid intolerable adverse reactions, a flexible dosing schedule will be used. According to the literature, this should be an average dose of about 1.75 mg base/day but is expected to vary between individuals. In a pilot study, the mean dose of pramipexole among participants was 2.51 mg base/day (equivalent to 3.59 mg salt/day). For example, D3 receptors are known to vary with age (fewer at older ages) and thus older individuals tolerate and require higher doses to achieve treatment efficacy. Blood and cerebrospinal fluid (CSF) samples are taken for analysis of dopamine and inflammatory markers and for genetic analysis linked to these systems to investigate any association between inflammation and anhedonia symptoms, brain reward-system dysfunction and treatment response to pramipexole. In addition, an fMRI study (Monetary Incentive Delay task: reward-system test) is planned to be performed before and after treatment with pramipexole, which can be used in future follow-up studies to investigate reward-system dysfunction in anhedonia and for predictive analyses of the treatment effect of pramipexole.

Prior to the baseline visit, fMRI screening is performed for the research subjects participating in the fMRI sub-trial. Before the research subject starts treatment with pramipexole or placebo, blood samples (and CSF if the research subject is participating in the CSF sub-trial) will be taken for storage in a biobank. Study participants are assessed with Snaith-Hamilton Pleasure Scale, Hamilton Depression 6-item rating scale and self-assessed with Dimensional Anhedonia Rating Scale, Montgomery-Åsberg Depression Rating Scale, Apathy Evaluation Scale, Insomnia Severity Scale, Generalized Anxiety Disorder 7-item rating scale and Brunnsviken Brief Quality of Life scale. Trial drugs are dispensed by trial staff and the study participant begins treatment according to a titration schedule. A dosing diary is distributed and the research subject is instructed to bring this completed diary to the next visit. Activity measurement results between screening and baseline are noted and activity measurement continues while treatment with pramipexole is given. Before starting pramipexole treatment, an fMRI examination and lumbar puncture will be performed for the research subjects participating in the sub-trial(s).

After the screening visit and randomization, an unblinded staff member places the correct packs of either placebo or active treatment in different concentrations to be distributed during the study in a box unique to each research subject. A logbook is kept of the packages placed in each box. Study participants are given oral and written information on how to take the tablets. Every third week during the study, the research subject will be called for a physical visit to discuss symptom assessment, titration plan and adverse reactions (using rating scales): New estimates including SHAPS and HDRS-6 are performed. Monitoring of adverse reactions, such as the onset of mania and impulse control disorders such as gambling addiction, is carried out using a form based on the Young Ziegler Mania Rating Scale (YMRS), Problem Gambling Severity Index (PGSI) and Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease (QUIP). Compliance is assessed as sufficient for continued participation in the study. If intolerable adverse reactions develop, the research subject will be asked to contact the investigator and the strategy will be to return to the last tolerable dose and wait seven days before attempting a new dose increase. Activity meters will be checked at follow-up visits. At the time of the visit, the research subject receives investigational medicinal products until the next scheduled visit and information on how to take them. Unused medicines are collected for compliance checks. Dispensed and returned trial medicines are logged. Between visits, research subjects are contacted by telephone to check on their titration status and possible adverse reactions.

After nine weeks, a final visit is made. New blood samples for the biobank are taken at the time of the visit. New fMRI examination and lumbar puncture will be performed on the research subjects participating in the sub-trial. The maximum tolerable dose of pramipexole is noted and new psychometric estimates are performed. Activity meters are read and submitted. After completing the study, the research participant will see an unblinded doctor at the clinic. If the research subject is randomized to active treatment, they have a choice to either continue pramipexole (but outside of the trial) or to taper pramipexole according to the tapering schedule.

To be able to compare fMRI examination and biomarkers between depressed and healthy controls, 40 healthy controls will also be recruited. The healthy controls will undergo blood sampling, lumbar puncture and fMRI according to the same protocol as the depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 75 years.
* Informed consent
* Diagnosis of unipolar depressive episode or bipolar disorder in depressive phase or dysthymia.
* Clinically significant anhedonia symptoms: SHAPS self-report score 3 or 4 on ≥ 3 items.
* Ongoing stable treatment with at least one antidepressant or mood stabilizing medication for at least 4 weeks. Has tried an antidepressant at a therapeutic dose but not achieved remission (refractory stage 1 depression)

Exclusion Criteria:

* Ongoing pregnancy, breastfeeding or planned pregnancy.
* High risk of suicide according to the overall clinical assessment of the research physician.
* Substance abuse within the last 6 months.
* Diagnosis of current psychotic disorder.
* Known diagnosis of Emotionally unstable personality disorder.
* Ongoing treatment under the Compulsory Psychiatric Care Act.
* Medical history or strong clinical suspicion of impulse control disorder (including current binge-eating disorder) or a current Attention Deficit Hyperactivity Disorder diagnosis with hyperactivity.
* Diagnosis of intellectual disability, dementia, or other circumstances that makes it difficult to understand the meaning of participating in the trial and provide informed consent.
* Diagnosis of renal failure (eGFR < 50 ml/min/1.73m2) or severe cardiovascular disease (specifically symptomatic heart failure New York Heart Association Class II or greater).
* Recently started psychotherapy (within 6 weeks) or planning to start such treatment during participation in the trial.
* Ongoing treatment with electroconvulsive therapy (ECT), ketamine or repetitive transcranial magnetic stimulation (rTMS), except maintenance ECT, ketamine or rTMS. (Maintenance treatment is defined as the use of ECT/ketamine/rTMS for a period exceeding 3 months after a series of ECT/ketamine/rTMS treatment in order to prevent the onset of a new episode.
* Other medical conditions or other concomitant drug treatment which, in the opinion of the investigators, may affect the evaluability of the trial or conditions that increase trial risk. For example, Parkinson's disease, hepatic insufficiency, ongoing cancer not in remission for more than one year, obesity surgery affecting the absorption of extended-release tablets.
* Ongoing treatment with drugs that affect plasma levels of pramipexole or have similar or antagonistic mechanism of action as pramipexole are not allowed. Ongoing treatment with neuroleptics are not allowed except for low-dose quetiapine 27 (≤150 mg/day) since it has very low binding to dopamine receptors at such low doses.
* Known or suspected allergy to any active substance or excipient in the medicinal product included in the trial.
* Participation in other treatment studies
* Other reason, as assessed by the investigator, that prevents the research subject's participation, such as the risk that the research subject is unable to complete the trial (non-compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Effect on anhedonia symptoms | 9 weeks
  Change in Snaith-Hamilton Pleasure Scale (SHAPS) self-report total score from baseline to week 9. Higher scores equal more severe anhedonoa. Score range 14-56

SECONDARY OUTCOMES:
Effect on core depression symptoms | 9 weeks
  Change in Hamilton Rating Scale for Depression 6 items (HDRS-6) total score baseline to week 9
Effect on other anhedonic domains not measured by SHAPS | 9 weeks
  Change in Dimensional Anhedonia Rating Scale (DARS) total score (inverse scale, lower points equals more anhedonia) from baseline to week 9
Effect on general depressive symptoms | 9 weeks
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS-S) total score from baseline to week 9
Effect on sleep disturbances | 9 weeks
  Change in Insomnia Severity Index (ISI) total score from baseline to week 9
Effect on apathy symptoms | 9 weeks
  Change in Apathy Evaluation Scale (AES) total score from baseline to week 9
Effect on anxiety symptoms | 9 weeks
  Change in Generalized Anxiety Disorder 7-item scale (GAD-7) total score from baseline to week 9
Effect on quality of life | 9 weeks
  Change in Brunnsviken Brief Quality of life scale (BBQ) total score from baseline to week 9
Effect on number of steps | 9 weeks
  Change in parameter "number of steps" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on distance travelled | 9 weeks
  Change in parameter "distance travelled" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on distribution of movement pattern over the day | 9 weeks
  Change in parameter "distribution of movement pattern over the day" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on sedantary behaviour | 9 weeks
  Change in parameter "sedentary behaviour" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on time spent in light | 9 weeks
  Change in parameter "time spent in light" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on moderate and vigorous physical activity | 9 weeks
  Change in parameter "moderate and vigorous physical activity" measured with a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on sleep latency | 9 weeks
  Change in parameter sleep latency (= time to fall asleep) using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on sleep awakening | 9 weeks
  Change in parameter sleep awakening (= how often one wakes up during the night) using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on wakefulness | 9 weeks
  Change in parameter wakefulness (=time in minutes awake during one night) using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on time in deep sleep | 9 weeks
  Change in parameter "time in deep sleep" using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on movement during sleep cycles | 9 weeks
  Change in parameter "movement during sleep cycles" using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Effect on sleep efficiency | 9 weeks
  Change in parameter sleep efficiency (=sleep time vs total time spent in bed) using a digital activity monitor (accelerometry bracelet), from baseline to week 9
Adverse events | 9 weeks
  Number and severity of adverse events
Effect on task-based brain signal variability in the reward circuit | 9 weeks
  BOLD-signaling during functional magnetic resonance imaging (fMRI) with Monetary Incentive Delay (MID)-task measuring Blood-Oxygen Level Dependent (BOLD) imaging pre/post treatment: Change in BOLD signals in nucleus accumbens from baseline to week 9
L-DOPA, blood: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of L-DOPA in blood sample from baseline to week 9
L-DOPA, CSF: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of L-DOPA in cerebrospinal fluid sample from baseline to week 9
Homovanillic acid, blood: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of homovanillic acid in blood sample from baseline to week 9
Homovanillic acid, CSF: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of homovanillic acid in cerebrospinal fluid sample from baseline to week 9
BH4, blood: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of tetrahydrobiopterin (BH4) in blood sample from baseline to week 9
BH4, CSF: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of tetrahydrobiopterin (BH4) in cerebrospinal fluid sample from baseline to week 9
Tyrosine, blood: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of tyrosine in blood sample from baseline to week 9
Tyrosine, CSF: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of tyrosine in cerebrospinal fluid sample from baseline to week 9
Phenylalanine, blood: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of phenylalanine in blood sample from baseline to week 9
Phenylalanine, CSF: biomarker of dopaminergic neurotransmission | 9 weeks
  Change in levels of phenylalanine in cerebrospinal fluid sample from baseline to week 9
IL-6, blood: biomarker of inflammation | 9 weeks
  Change in levels of interleukin-6 (IL-6) in blood sample from baseline to week 9
IL-6, CSF: biomarker of inflammation | 9 weeks
  Change in levels of interleukin-6 (IL-6) in cerebrospinal fluid sample from baseline to week 9
IL-1b, blood: biomarker of inflammation | 9 weeks
  Change in levels of interleukin-1b (IL-1b) in blood sample from baseline to week 9
IL-1b, CSF: biomarker of inflammation | 9 weeks
  Change in levels of interleukin-1b (IL-1b) in cerebrospinal fluid sample from baseline to week 9
IFN-y, blood: biomarker of inflammation | 9 weeks
  Change in levels of interferon gamma (IFN-y) in blood sample from baseline to week 9
IFN-y, CSF: fluid biomarker of inflammation | 9 weeks
  Change in levels of interferon gamma (IFN-y) in cerebrospinal fluid sample from baseline to week 9
hs-CRP, blood: biomarker of inflammation | 9 weeks
  Change in levels of high-sensitivity C-reactive peptide (hs-CRP) in blood sample from baseline to week 9
hs-CRP, CSF: biomarker of inflammation | 9 weeks
  Change in levels of high-sensitivity C-reactive peptide (hs-CRP) in cerebrospinal fluid from baseline to week 9
TNF, blood: biomarker of inflammation | 9 weeks
  Change in levels of tumor necrosis factor-alpha (TNF-alpha) in blood sample from baseline to week 9
TNF, CSF: biomarker of inflammation | 9 weeks
  Change in levels of tumor necrosis factor-alpha (TNF-alpha) in cerebrospinal fluid from baseline to week 9
Cognitive function pre/post Treatment | 9 weeks
  Change in cognitive performance using the WAIS-IV
Cognitive function pre/post Treatment | 9 weeks
  Change in cognitive performance using the Repeatable Battery for the Assessment of Neuropsychological Status.
Cognitive function pre/post Treatment | 9 weeks
  Change in cognitive performance using the Delis-Kaplan Executive Function System.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindahl J, Asp M, Stahl D, Tjernberg J, Eklund M, Bjorkstrand J, van Westen D, Jensen J, Mansson K, Tornberg A, Svensson M, Deierborg T, Ventorp F, Lindqvist D. Add-on pramipexole for anhedonic depression: study protocol for a randomised controlled trial and open-label follow-up in Lund, Sweden. BMJ Open. 2023 Nov 30;13(11):e076900. doi: 10.1136/bmjopen-2023-076900. PMID 38035737

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT05355337/SAP_000.pdf